CLINICAL TRIAL: NCT03574090
Title: PROTOP: Study of the Efficacy of Topical Antibiotherapy in the Prophylaxis of Incisional Surgical Localization Infection in Colorectal Surgery
Brief Title: Study the Efficacy of Topical Antibiotherapy in the Prophylaxis of Incisional Surgical Infection in Colorectal Surgery
Acronym: PROTOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Miquel Casal Rossell, General Surgeon, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1234
Record Dates: First submitted 2018-05-30; First posted 2018-06-29 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Surgical Wound Infection; Postoperative Wound Infection; Postoperative Wound Infection Superficial Incisional; Preventive Therapy
Keywords: topical antibiotic; surgical wound infection; prevention of surgical wound infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Amoxicillin-Potassium Clavulanate Combination; Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In the operating room area we will keep a notebook with the random number sheet and a box with the numbered envelopes and containing the treatment to follow: physiological saline alone or physiological saline with antibiotic. At the end of the surgery and before closing the abdominal wall, it is definitively informed to the nurse whether or not to recruit them, a case number is assigned chronologically and in the random number sheet corresponds to an envelope containing one of the two treatments. Dilution is performed with 10cc of physiological saline solution with or without antibiotic in the outside of the operating room and then it is incorporated into the 500cc bottle of physiological saline once opened in a sterile way. We used according to the usual protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amoxicillin clavulanate (Experimental): 1000 mg amoxicillin and potassium clavulanate equivalent to 200mg of clavulanic acid. administered topically and dissolved in 500 ml 0.9% Physiological Serum.
  Interventions: Drug: Amoxicillin Clavulanate; Drug: Physiological Saline
- Physiological Saline (Active Comparator): 500 milliliters of 0.9% Physiological Serum.
  Interventions: Drug: Physiological Saline

INTERVENTIONS:
Drug: Amoxicillin Clavulanate — To demonstrate its efficacy in the prophylaxis of infection to surgical wound will be used in dirty/contaminated emergency surgery and its efficacy will be compared with topical administration of physiological serum alone.
  Other Names: 1000 mg amoxicillin and 200mg clavulanic acid.
  Arms: amoxicillin clavulanate
Drug: Physiological Saline — To demonstrate its efficacy in the prophylaxis of infection to surgical wound will be used in dirty/contaminated emergency surgery and its efficacy will be compared with topical administration of physiological serum alone.
  Other Names: 500 milliliters of 0.9% Physiological Serum

SUMMARY:
The main objective is to study the efficacy of topical antibiotic therapy with Amoxicillin / Clavulanic acid in the prevention of surgical wound infection in patients undergoing to colorectal surgery

DETAILED DESCRIPTION:
Is a clinical trial phase IV prospective, blind, controlled and random allocation of treatment with the active principle of amoxicillin 1000mg and 200mg Clavulanic acid, administered topically and dissolved in 500 ml of saline 0.9%. To demonstrate its effectiveness in the surgical wound infection prophylaxis be used in contaminated surgery and be compared its effectiveness with the topical administration of normal saline only.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients who require urgent surgical intervention and who come from the emergency service
* Patients affected by complicated intra-abdominal infection with peritonitis of more than one abdominal compartment or intra-abdominal abscess requiring open surgical intervention.

Exclusion Criteria:

* Women patients with positive pregnancy test.
* Patients with primary peritonitis and liver cirrhosis.
* Patients who have received antibiotic treatment during the 72 hours prior to the surgical intervention (except that administered to UCIES as a treatment dose of the same process)
* Patients allergic to the antibiotic used in the study.
* Patients who have undergone a surgical procedure of recently opened abdomen (up to 30 days before surgery), a prosthesis of synthetic material (mesh) or to which the surgical wound can not be closed according to the surgeon's criteria.
* Patients with an unfavorable life prognosis (ASA 5).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of topical antibiotic prophylaxis on the incidence of SSI | 30 days
  Evaluation of the effect of topical antibiòtic ( Amoxicillin 1000mg and 200mg of Clavulanic acid dissolved in 500 milliliters of 0.9% Physiological Serum ) prophylaxis on the incidence of Surgical Site Infection in surgery due to emergency intra-abdominal infection

SECONDARY OUTCOMES:
reduction of hospital stay | 30 days
  Effect of the protocol of topical prophylaxis in the reduction of hospital stay
Bacterial charge | 30 days
  Effect of topical prophylaxis protocol on reducing bacterial charge
Bacterial resistance | 30 days
  Effect of topical prophylaxis protocol on Bacterial resistance

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Badia Perez, PH. D, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] National Nosocomial Infections Surveillance (NNIS) report, data summary from October 1986-April 1996, issued May 1996. A report from the National Nosocomial Infections Surveillance (NNIS) System. Am J Infect Control. 1996 Oct;24(5):380-8. No abstract available. PMID 8902113
- [Result] Anderson DJ, Sexton DJ, Kanafani ZA, Auten G, Kaye KS. Severe surgical site infection in community hospitals: epidemiology, key procedures, and the changing prevalence of methicillin-resistant Staphylococcus aureus. Infect Control Hosp Epidemiol. 2007 Sep;28(9):1047-53. doi: 10.1086/520731. Epub 2007 Jul 12. PMID 17932825
- [Result] Simmons BP. Cdc guidelines on infection control. Infect Control. 1982 Mar-Apr;3(2 Suppl):187-96. doi: 10.1017/s0195941700056721. No abstract available. PMID 6918373
- [Result] Charalambous CP, Tryfonidis M, Swindell R, Lipsett AP. When should old therapies be abandoned? A modern look at old studies on topical ampicillin. J Infect. 2003 Oct;47(3):203-9. doi: 10.1016/s0163-4453(03)00071-9. PMID 12963381
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Chura JC, Boyd A, Argenta PA. Surgical site infections and supplemental perioperative oxygen in colorectal surgery patients: a systematic review. Surg Infect (Larchmt). 2007 Aug;8(4):455-61. doi: 10.1089/sur.2006.034. PMID 17883362
- [Result] Culver DH, Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG, Banerjee SN, Edwards JR, Tolson JS, Henderson TS, et al. Surgical wound infection rates by wound class, operative procedure, and patient risk index. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):152S-157S. doi: 10.1016/0002-9343(91)90361-z. PMID 1656747
- [Result] Friberg O, Svedjeholm R, Soderquist B, Granfeldt H, Vikerfors T, Kallman J. Local gentamicin reduces sternal wound infections after cardiac surgery: a randomized controlled trial. Ann Thorac Surg. 2005 Jan;79(1):153-61; discussion 161-2. doi: 10.1016/j.athoracsur.2004.06.043. PMID 15620935
- [Result] Lazar HL, Ketchedjian A, Haime M, Karlson K, Cabral H. Topical vancomycin in combination with perioperative antibiotics and tight glycemic control helps to eliminate sternal wound infections. J Thorac Cardiovasc Surg. 2014 Sep;148(3):1035-8; 1038-40. doi: 10.1016/j.jtcvs.2014.06.045. Epub 2014 Jul 2. PMID 25129595
- [Result] Garner JS. CDC guideline for prevention of surgical wound infections, 1985. Supersedes guideline for prevention of surgical wound infections published in 1982. (Originally published in November 1985). Revised. Infect Control. 1986 Mar;7(3):193-200. doi: 10.1017/s0195941700064080. No abstract available. PMID 3633903
- [Result] Abdullah KG, Attiah MA, Olsen AS, Richardson A, Lucas TH. Reducing surgical site infections following craniotomy: examination of the use of topical vancomycin. J Neurosurg. 2015 Dec;123(6):1600-4. doi: 10.3171/2014.12.JNS142092. Epub 2015 Jun 19. PMID 26090835
- [Result] Kang DG, Holekamp TF, Wagner SC, Lehman RA Jr. Intrasite vancomycin powder for the prevention of surgical site infection in spine surgery: a systematic literature review. Spine J. 2015 Apr 1;15(4):762-70. doi: 10.1016/j.spinee.2015.01.030. Epub 2015 Jan 28. PMID 25637469
- [Result] Kirby JP, Mazuski JE. Prevention of surgical site infection. Surg Clin North Am. 2009 Apr;89(2):365-89, viii. doi: 10.1016/j.suc.2009.01.001. PMID 19281889
- [Result] Krukowski ZH, Irwin ST, Denholm S, Matheson NA. Preventing wound infection after appendicectomy: a review. Br J Surg. 1988 Oct;75(10):1023-33. doi: 10.1002/bjs.1800751023. PMID 3064867
- [Result] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Result] Musters GD, Burger JW, Buskens CJ, Bemelman WA, Tanis PJ. Local Application of Gentamicin in the Prophylaxis of Perineal Wound Infection After Abdominoperineal Resection: A Systematic Review. World J Surg. 2015 Nov;39(11):2786-94. doi: 10.1007/s00268-015-3159-5. PMID 26170157
- [Result] Leaper D, Burman-Roy S, Palanca A, Cullen K, Worster D, Gautam-Aitken E, Whittle M; Guideline Development Group. Prevention and treatment of surgical site infection: summary of NICE guidance. BMJ. 2008 Oct 28;337:a1924. doi: 10.1136/bmj.a1924. No abstract available. PMID 18957455
- [Result] Rutten HJ, Nijhuis PH. Prevention of wound infection in elective colorectal surgery by local application of a gentamicin-containing collagen sponge. Eur J Surg Suppl. 1997;(578):31-5. PMID 9167147
- [Result] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Result] Nichols RL. Preventing surgical site infections: a surgeon's perspective. Emerg Infect Dis. 2001 Mar-Apr;7(2):220-4. doi: 10.3201/eid0702.010214. PMID 11294711
- [Result] Serrano-Heranz R. [Antimicrobial prophylaxis for surgery]. Rev Esp Quimioter. 2006 Dec;19(4):323-31. No abstract available. Spanish. PMID 17235400
- [Result] Rosen HR, Marczell AP, Czerwenka E, Stierer MO, Spoula H, Wasl H. Local gentamicin application for perineal wound healing following abdominoperineal rectum excision. Am J Surg. 1991 Nov;162(5):438-41. doi: 10.1016/0002-9610(91)90256-d. PMID 1951905
- [Result] Schultz A, Jorgensen PM, Jorgensen SP. Septic complications after appendicectomy for perforated appendicitis. A controlled clinical trial metronidazole and topical ampicillin. Acta Chir Scand. 1983;149(5):517-20. PMID 6356732
- [Result] Sessler DI, Akca O. Nonpharmacological prevention of surgical wound infections. Clin Infect Dis. 2002 Dec 1;35(11):1397-404. doi: 10.1086/344275. Epub 2002 Nov 13. PMID 12439804
- [Result] Tweed C. Prevention of surgical wound infection: prophylactic antibiotics in colorectal surgery. J Wound Care. 2005 May;14(5):202-5. doi: 10.12968/jowc.2005.14.5.26769. PMID 15909433
- [Result] Sociedad Española de Medicina Preventiva, Salud Pública e Higiene (SEMPSPH). (2015). Evolución EPINE 1990-2015 de la prevalencia de las infecciones nosocomiales en los hospitales españoles. EPINE. 1990-2015. Madrid.
- [Result] Vasavada AR, Gajjar D, Raj SM, Vasavada V, Vasavada V. Comparison of 2 moxifloxacin regimens for preoperative prophylaxis: prospective randomized triple-masked trial. Part 1: aqueous concentration of moxifloxacin. J Cataract Refract Surg. 2008 Aug;34(8):1379-82. doi: 10.1016/j.jcrs.2008.04.027. PMID 18655991
- [Result] Wilson AP, Treasure T, Sturridge MF, Gruneberg RN. A scoring method (ASEPSIS) for postoperative wound infections for use in clinical trials of antibiotic prophylaxis. Lancet. 1986 Feb 8;1(8476):311-3. doi: 10.1016/s0140-6736(86)90838-x. PMID 2868173
- [Result] X.Guirao, J. A. (2006). Infecciones quirúrgicas (Guías clínicas de la asociación española de cirujanos).
- [Result] Yan H, He J, Chen S, Yu S, Fan C. Intrawound application of vancomycin reduces wound infection after open release of post-traumatic stiff elbows: a retrospective comparative study. J Shoulder Elbow Surg. 2014 May;23(5):686-92. doi: 10.1016/j.jse.2014.01.049. PMID 24745317
- [Result] Badia JM, Martinez-Rodenas F, Oms LM, Valverde J, Franch G, Rosales A, Serrano R, Sitges-Serra A. [A randomized prospective study of antibiotic prophylaxis compared to lavage of the surgical wound in nonperforating appendicitis]. Med Clin (Barc). 1994 Jul 9;103(6):201-4. Spanish. PMID 7967862
- [Result] Badia JM, de la Torre R, Farre M, Gaya R, Martinez-Rodenas F, Sancho JJ, Sitges-Serra A. Inadequate levels of metronidazole in subcutaneous fat after standard prophylaxis. Br J Surg. 1995 Apr;82(4):479-82. doi: 10.1002/bjs.1800820417. PMID 7613890
- [Result] Badia JM, Torres JM, Tur C, Sitges-Serra A. Saline wound irrigation reduces the postoperative infection rate in guinea pigs. J Surg Res. 1996 Jul 1;63(2):457-9. doi: 10.1006/jsre.1996.0292. PMID 8661242
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Badia JM, Del Toro MD, Navarro Gracia JF, Balibrea JM, Herruzo R, Gonzalez Sanchez C, Lozano Garcia J, Rubio Perez I, Guirao X, Soria-Aledo V, Orti-Lucas R; Surgical Location Infection Prevention Program Working Group of the Observatory of Infection in Surgery. Surgical Infection Reduction Program of the Observatory of Surgical Infection (PRIQ-O): Delphi prioritization and consensus document on recommendations for the prevention of surgical site infection. Cir Esp (Engl Ed). 2023 Apr;101(4):238-251. doi: 10.1016/j.cireng.2022.11.009. Epub 2022 Nov 24. PMID 36427782
- [Result] Foschi D, Yakushkina A, Cammarata F, Lamperti G, Colombo F, Rimoldi S, Antinori S, Sampietro GM. Surgical site infections caused by multi-drug resistant organisms: a case-control study in general surgery. Updates Surg. 2022 Oct;74(5):1763-1771. doi: 10.1007/s13304-022-01243-3. Epub 2022 Mar 19. PMID 35304900
- [Result] Gomes ET, Carbogim FDC, Lins RS, Lins-Filho RLM, Poveda VB, Puschel VAA. Effectiveness of supplemental oxygenation to prevent surgical site infections: A systematic review with meta-analysis. Rev Lat Am Enfermagem. 2022 Oct 7;30:e3648. doi: 10.1590/1518-8345.6106.3648. eCollection 2022. PMID 36228236
- [Result] Arroyo-Garcia N, Badia JM, Vazquez A, Pera M, Pares D, Limon E, Almendral A, Piriz M, Diez C, Fraccalvieri D, Lopez-Contreras J, Pujol M; Members of the VINCat Colorectal Surveillance Team; VINCat Program. An interventional nationwide surveillance program lowers postoperative infection rates in elective colorectal surgery. A cohort study (2008-2019). Int J Surg. 2022 Jun;102:106611. doi: 10.1016/j.ijsu.2022.106611. Epub 2022 Apr 12. PMID 35427799
- [Result] Fuglestad MA, Tracey EL, Leinicke JA. Evidence-based Prevention of Surgical Site Infection. Surg Clin North Am. 2021 Dec;101(6):951-966. doi: 10.1016/j.suc.2021.05.027. PMID 34774274
- [Result] Chen S, Chen JW, Guo B, Xu CC. Preoperative Antisepsis with Chlorhexidine Versus Povidone-Iodine for the Prevention of Surgical Site Infection: a Systematic Review and Meta-analysis. World J Surg. 2020 May;44(5):1412-1424. doi: 10.1007/s00268-020-05384-7. PMID 31996985
- [Result] Badia JM, Casey AL, Rubio-Perez I, Arroyo-Garcia N, Espin E, Biondo S, Balibrea JM. Awareness of Practice and Comparison with Best Evidence in Surgical Site Infection Prevention in Colorectal Surgery. Surg Infect (Larchmt). 2020 Apr;21(3):218-226. doi: 10.1089/sur.2019.203. Epub 2019 Nov 14. PMID 31724910
- [Result] Badia JM, Casey AL, Rubio-Perez I, Crosby C, Arroyo-Garcia N, Balibrea JM. A survey to identify the breach between evidence and practice in the prevention of surgical infection: Time to take action. Int J Surg. 2018 Jun;54(Pt A):290-297. doi: 10.1016/j.ijsu.2018.04.038. Epub 2018 Apr 25. PMID 29704562
- [Result] Kamboj M, Childers T, Sugalski J, Antonelli D, Bingener-Casey J, Cannon J, Cluff K, Davis KA, Dellinger EP, Dowdy SC, Duncan K, Fedderson J, Glasgow R, Hall B, Hirsch M, Hutter M, Kimbro L, Kuvshinoff B, Makary M, Morris M, Nehring S, Ramamoorthy S, Scott R, Sovel M, Strong V, Webster A, Wick E, Aguilar JG, Carlson R, Sepkowitz K. Risk of Surgical Site Infection (SSI) following Colorectal Resection Is Higher in Patients With Disseminated Cancer: An NCCN Member Cohort Study. Infect Control Hosp Epidemiol. 2018 May;39(5):555-562. doi: 10.1017/ice.2018.40. Epub 2018 Mar 19. PMID 29553001
- [Result] Farach SM, Kelly KN, Farkas RL, Ruan DT, Matroniano A, Linehan DC, Moalem J. Have Recent Modifications of Operating Room Attire Policies Decreased Surgical Site Infections? An American College of Surgeons NSQIP Review of 6,517 Patients. J Am Coll Surg. 2018 May;226(5):804-813. doi: 10.1016/j.jamcollsurg.2018.01.005. Epub 2018 Feb 28. PMID 29408507
- [Result] Pieper D, Rombey T, Doerner J, Rembe JD, Zirngibl H, Zarras K, Ambe PC. The role of saline irrigation prior to wound closure in the reduction of surgical site infection: protocol for a systematic review and meta-analysis. Syst Rev. 2018 Oct 5;7(1):152. doi: 10.1186/s13643-018-0813-7. PMID 30286812
- [Result] Nelson RL, Iqbal NM, Kravets A, Khateeb R, Raza M, Siddiqui M, Taha I, Tummala A, Epple R, Huang S, Wen M. Topical antimicrobial prophylaxis in colorectal surgery for the prevention of surgical wound infection: a systematic review and meta-analysis. Tech Coloproctol. 2018 Aug;22(8):573-587. doi: 10.1007/s10151-018-1814-1. Epub 2018 Jul 17. PMID 30019145
- See also: VINCat — https://catsalut.gencat.cat/ca/proveidors-professionals/vincat/
- See also: health prevention — https://scientiasalut.gencat.cat/handle/11351/3304